CLINICAL TRIAL: NCT05615519
Title: Validation of a Smartphone-based Intelligent Diagnosis and Measurement for Strabismus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Other Study IDs: DRStrabismus2022
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Strabismus; Exotropia; Esotropia; Vertical Strabismus
Keywords: Mobile health; Artificaial intelligence medicine; Pediatric ophthalmology
MeSH Terms: conditions — Strabismus; Exotropia; Esotropia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eligible participants for smartphone-based strabismus measurement and diagnosis: Facial videos dataset Facial videos were collected using smartphone and following the programmatic cover tests.
  Interventions: Diagnostic Test: A new technology based on 3D reconstruction and deep learning algorithm to achieve an automatic diagnosis of strabismus based on patient-sourced videos of programmatic cover tests.

INTERVENTIONS:
Diagnostic Test: A new technology based on 3D reconstruction and deep learning algorithm to achieve an automatic diagnosis of strabismus based on patient-sourced videos of programmatic cover tests. — Digital ruler of strabismus

SUMMARY:
The current measurement methods of strabismus include the corneal light reflection method, prism alternate covering, etc., which especially rely on the subjective experience of doctors, and there is a large error between different measurers， leading to serious underestimation of strabismus prevalence and insufficient care for strabismus patients. Here, the investigators established and validated an artificial intelligence system to achieve an automatic diagnosis of strabismus based on patient-sourced videos of programmatic cover tests. Three-dimensional reconstruction methods are used to digitize the parameters of head and eye positions. This system has been integrated into a smartphone platform to be further validated through hospital-based and population-based clinical trials.

ELIGIBILITY:
Inclusion Criteria:

The quality of facial videos should be clinically acceptable.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients from strabismus & optometry departments or participants from the internet.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-12-02 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of smartphone-based diagnosis | Baseline
  The accurate and the area under curve of the smartphone-based diagnosis.
The consistency between manual and smartphone measurement | Baseline
  Agreement between the manual and automated tests was represented in Bland-Altman plots and concordance correlation coefficients.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity, Guangzhou, Guangdong, China